CLINICAL TRIAL: NCT02032693
Title: The Effect of Dietary Supplementation on DNA Damage, Inflammation, Stress, and Related Factors Important in Somatic and Stem Cell Senescence in Healthy Adults
Brief Title: Everycell's Effect on DNA Damage, Inflammation, and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: CellHealth Institute (Unknown)
Responsible Party: Principal Investigator, John E. Lewis, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20130411
Record Dates: First submitted 2014-01-02; First posted 2014-01-10 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Family Member
Keywords: Everycell; DNA damage; DNA inflammation; DNA stress
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everycell™ (Experimental): Patient will take 1 tablet two times daily of Everycell™ (double-blind) for the 4-week treatment period.
  Interventions: Dietary Supplement: Everycell™
- Placebo (Placebo Comparator): Patient will take 1 tablet two times daily of the placebo (double-blind) for the 4-week treatment period.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Everycell™
  Arms: Everycell™
Other: Placebo
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The investigators are conducting this research because they want to determine if a dietary supplement, called Everycell™, has an effect on the functioning of the study participants' cells. The results of this research will be used to help develop additional strategies for trying to fight the effects of aging. The primary purpose of this study is to determine the effectiveness of Everycell™ compared to placebo (a pill that does nothing) on DNA damage, inflammation, stress, and related factors. Taking Everycell™ is not a medical prescription, treatment, or cure for any known disease or condition.

Helping patients' nutritional status is important to prevent the continued worsening of chronic diseases and also to counteract the effects of aging. Americans also have difficulties with compliance to prescription medications due to their toxicity and side effects. This study aims to learn more about how a dietary supplement may improve nutritional status and enable the body to normalize cellular functioning, which may improve quality of life. The results of this research will be used to determine if Everycell™ is beneficial for overall cellular health and to counteract the effects of aging.

DETAILED DESCRIPTION:
The proposed study is a 6-week, randomized, double-blind, placebo-controlled trial to evaluate the effect of everycell compared to placebo on DNA damage, inflammation, stress, and related factors in 30 healthy adults (18-55 years of age). Participants will be assessed at baseline, 4 weeks (end of intervention), and 6 weeks (2-week washout period), and the study will consist of two treatment arms, including: (a) Everycell and (b) placebo. Additionally, the study will examine subject health-related quality of life (QoL).

Specific Aim. Test the effect of Everycell compared to placebo on DNA damage, inflammation, stress, and related factors in a sample of healthy adults.

Hypothesis. The Everycell group will demonstrate improvements in DNA damage, inflammation, stress, and related factors at 4 and 6-week follow-ups compared to placebo.

Although all measures to protect confidentiality will be put in place, the possibility exists that electronic data could be jeopardized. In the remote case that such event occurs, it will be immediately reported to the IRB.

No substantial psychological, medical, or social risks exist to the participants, other than minor discomfort associated with the venipuncture. The components of everycell should be harmless without significant food allergies. No serious, untoward side effects have been reported to the company by consumers nor observed during previous human studies. If any side effect does occur, the remedy is to discontinue until asymptomatic, and then reintroduce at 1/4 dosage, increasing by the same amount every 2 days, if uneventful, until full dosage is achieved. A toxicology search for each component reveals no unique toxicity characteristic of the materials. As reported by CellHealth Institute, the manufacturer of the product, many customers currently use Everycell, and CellHealth Institute is unaware of significant toxicities.

CellHealth Institute applies the latest scientific methods to ensure the value and safety of their raw materials. CellHealth Institute products are manufactured in state-of-the-art facilities, under strict quality control and environmental protection standards.

Participants will incur no additional appreciable psychological or social risks by participating in this study, although they may undergo psychological and physical discomfort sometimes. The process of interviewing during the assessment may cause discomfort. Discomfort or fatigue may also be experienced in completing the assessment battery.

Alternatives to this study for improving DNA damage, inflammation, and stress include prescription medications, exercise, dietary modification, and other nutritional supplements. The risks of medications can be very significant, including life-threatening, but the risk of taking nutritional supplements is not totally understood, since they are not regulated by the US Food and Drug Administration. Medications and nutritional supplements, as part of a change in lifestyle behaviors, may also prove to be beneficial for DNA damage, inflammation, and stress, but their long-term use has unknown consequences.

The information obtained in this study will help in determining the efficacy of using a nutritional supplement for improving DNA damage, inflammation, and stress outcomes. By participating in the study, subjects may experience improved DNA damage, inflammation, and stress. The risk of participating in this study is reasonable because of the potential enhancements in DNA damage, inflammation, and stress with improved nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 55
* Live independently without medical assistance
* Willing to provide informed consent to participate in the study
* Willing to follow our procedures and requirements for the study, including:

  1. providing blood, urine, and saliva samples
  2. completing other assessments
* Patients may take a similar dietary supplement as the one used in the study, but they must stop taking all similar dietary supplements 2 weeks prior to starting the study and for the 6 weeks duration of the study.

Exclusion Criteria:

* Patients need to be free of major medical conditions, such as neurological, cardiovascular, pulmonary, renal, endocrine, thyroid, hepatic, autoimmune, or bone/joint disorders or conditions; psychiatric diagnoses or psychotic disorders, and have no gastrointestinal disorders that could affect how the dietary supplement is absorbed by their body.
* Cannot participate in another similar research trial within 30 days of participating in this study
* Cannot be a smoker or have stopped smoking less than 6 months ago
* Cannot currently be taking any chemotherapy or radiation treatment for cancer
* Cannot be diagnosed with a terminal illness
* Cannot be diagnosed with insulin-dependent diabetes and/or be taking metformin
* Cannot be HIV positive
* If female, the patient cannot currently be pregnant, breastfeeding, or intending to become pregnant within the next month

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Nuclear factor kappa-light-chain-enhancer of activated B cells at 4 weeks | Baseline, 4-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Fructosamine at 4 weeks | Baseline, 4-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Protein Thiol Test at 4 weeks | Baseline, 4-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Homocysteine at 4 weeks | Baseline, 4-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Telomere Length at 4 weeks | Baseline, 4-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Cluster of Differentiation 4 (Regulatory T-cell) at 4 weeks | Baseline, 4-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Cluster of Differentiation 8 at 4 weeks | Baseline, 4-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Cluster of Differentiation 56 (Natural Killer cell) at 4 weeks | Baseline, 4-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in 8-hydroxydeoxyguanosine at 4 weeks | Baseline, 4-week follow-up
  Urine sample for 8-OHdG and 8-epi-PGF-2-alpha
Change from Baseline in 8-epi-PGF-2-alpha at 4 weeks | Baseline, 4-week follow-up
  Urine sample for 8-OHdG and 8-epi-PGF-2-alpha
Change from Baseline in Forkhead box protein 3 (Regulatory T-cell) at 4 weeks | Baseline, 4-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Nuclear factor kappa-light-chain-enhancer of activated B cells at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Fructosamine at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Protein Thiol Test at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Homocysteine at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Telomere Length at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Cluster of Differentiation 4 (Regulatory T-cell) at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Cluster of Differentiation 8 at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Cluster of Differentiation 56 (Natural Killer cell) at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in 8-hydroxydeoxyguanosine at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in 8-epi-PGF-2-alpha at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)
Change from Baseline in Forkhead box protein 3 (Regulatory T-cell) at 6 weeks | Baseline, 6-week follow-up
  Blood draw for NF-kB, fructosamine, protein thiol test, homocysteine, telomere length, and CD4/FoxP3 (regulatory T-cells), CD8, and CD56 (NK cell)

SECONDARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure at 4 weeks | Baseline, 4-week follow-up
  Systolic and diastolic blood pressure measured.
Change from Baseline in Pulse at 4 weeks | Baseline, 4-week follow-up
Change from Baseline in Waist Circumference at 4 weeks | Baseline, 4-week follow-up
  Measure of body composition: waist circumference (cm).
Change from Baseline in Hip Circumference at 4 weeks | Baseline, 4-week follow-up
  Measure of body composition: hip circumference (cm).
Change from Baseline in Weight at 4 weeks | Baseline, 4-week follow-up
  Measure of body composition: weight.
Change from Baseline in Height at 4 weeks | Baseline, 4-week follow-up
  Measure of body composition: height.
Change from Baseline in Body Mass Index at 4 weeks | Baseline, 4-week follow-up
  Measure of body composition: height and weight to assess BMI.
Change from Baseline in International Physical Activity Questionnaire at 4 weeks | Baseline, 4-week follow-up
Change from Baseline in SF-36v2™ Health Survey at 4 weeks | Baseline, 4-week follow-up
Change from Baseline in Systolic Blood Pressure at 6 weeks | Baseline, 6-week follow-up
  Systolic and diastolic blood pressure measured.
Change from Baseline in Diastolic Blood Pressure at 4 weeks | Baseline, 4-week follow-up
  Systolic and diastolic blood pressure measured.
Change from Baseline in Diastolic Blood Pressure at 6 weeks | Baseline, 6-week follow-up
  Systolic and diastolic blood pressure measured.
Change from Baseline in Pulse at 6 weeks | Baseline, 6-week follow-up
Change from Baseline in Waist Circumference at 6 weeks | Baseline, 6-week follow-up
  Measure of body composition: waist circumference (cm).
Change from Baseline in Hip Circumference at 6 weeks | Baseline, 6-week follow-up
  Measure of body composition: hip circumference (cm).
Change from Baseline in Weight at 6 weeks | Baseline, 6-week follow-up
  Measure of body composition: weight.
Change from Baseline in Height at 6 weeks | Baseline, 6-week follow-up
  Measure of body composition: height.
Change from Baseline in Body Mass Index at 6 weeks | Baseline, 6-week follow-up
  Measure of body composition: height and weight to assess BMI.
Change from Baseline in International Physical Activity Questionnaire at 6 weeks | Baseline, 6-week follow-up
Change from Baseline in SF-36v2™ Health Survey at 6 weeks | Baseline, 6-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: John Lewis, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Clinical Research Building, Miami, Florida, United States